CLINICAL TRIAL: NCT06347029
Title: Evaluation of Endothelial Dysfunction Using the "Flow Mediated Dilation" Test in a Population of Chronic Renal Failure Patients at Different Stages, and Evaluation of the Role of Antiphospholipid Antibodies - A Prospective Interventional Study.
Brief Title: Evaluation of Endothelial Dysfunction Using the "Flow Mediated Dilation" Test in a Population of Chronic Renal Failure Patients at Different Stages, and Evaluation of the Role of Antiphospholipid Antibodies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Besse-Hammer, Head of clinical trial unit, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Endothelial dysfunction
Record Dates: First submitted 2024-03-25; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Chronic kidney disease at stage G3a (Experimental): Renal clearance according to CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) between 60 and 45 ml/min/1.73m²
  Interventions: Procedure: Urine sampling; Procedure: Blood sampling; Device: Flow mediated dilatation test
- Chronic kidney disease at stage G3b (Experimental): Renal clearance according to CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) between 45 and 30 ml/min/1.73m²
  Interventions: Procedure: Urine sampling; Procedure: Blood sampling; Device: Flow mediated dilatation test
- Chronic kidney disease at stage G4 (Experimental): Renal clearance according to CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) between 30 and 15 ml/min/1.73m²
  Interventions: Procedure: Urine sampling; Procedure: Blood sampling; Device: Flow mediated dilatation test
- Chronic kidney disease at stage G5 not dialyzed (Experimental): Renal clearance according to CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) less than 15 ml/min/1.73m² but not dialyzed
  Interventions: Procedure: Urine sampling; Procedure: Blood sampling; Device: Flow mediated dilatation test
- Chronic kidney disease at stage G5 with dialyze (Experimental): Patients who undergo dialyze
  Interventions: Procedure: Urine sampling; Procedure: Blood sampling; Device: Flow mediated dilatation test
- Control (Active Comparator): Healthy volunteer patient, without existing kidney disease
  Interventions: Procedure: Urine sampling; Procedure: Blood sampling; Device: Flow mediated dilatation test

INTERVENTIONS:
Procedure: Urine sampling — Urine sampling
Procedure: Blood sampling — Blood sampling
Device: Flow mediated dilatation test — The flow mediated dilation (FMD) test is the most commonly utilized, non-invasive, ultrasound assessment of endothelial function in humans.

SUMMARY:
The vascular endothelium is an organ in its own right, playing, among other things, a primordial role in the control of vascular tone. This vascular tone is ensured by pro-dilator mediators (nitric oxide (NO), prostacyclins (PGI2)), or vasoconstrictors (endothelin, thromboxane A2 or PGH2).Uremic toxin accumulation in chronic kidney disease (CKD) is a well-known factor in endothelial dysfunction, often associated with higher cardiovascular risk. This association is also present for terminal chronic kidney disease characterized by the need to resort to an extra-renal purification technique (in-center hemodialysis (HD), daily home hemodialysis (HDQ), peritoneal dialysis) or to resort to renal transplantation.

For HD to be effective, it is essential that the blood flow rate passing through the dialyzer is greater than 300ml/min. This imperative requires that any hemodialysis patient have specific vascular access (dialysis catheter or arteriovenous fistula (AVF)) to ensure these flow rates. The vascular access of choice is the arteriovenous fistula , because it is associated with a lower risk of infection and lower morbidity and mortality. Making an arteriovenous fistula consists of surgically creating an anastomosis between a vein and an artery.

Complications of arteriovenous fistula are common. Arteriovenous fistula maturation may be delayed (maturation delay) or even absent. Drainage veins and/or anastomoses can also be the site of stenosis or thrombosis. The pathophysiology of these complications is complex and multifactorial. Among the risk factors for these complications (delay or absence of maturation, stenosis thrombosis), the positivity of antiphospholipid antibodies (aPL) can be cited, as well as endothelial dysfunction.

Antiphospholipid syndrome (APS) is an autoimmune disease causing a thrombotic phenotype. This is an acquired thrombophilia. In the general population, the prevalence of antiphospholipid antibodies is around 0.5%; this prevalence is far from rare in hemodialysis, since it represents up to 37% in dialysis patients. In a retrospective study carried out at Brugmann University Hospital in 2023 , on 115 patients with AVF and in whom aPL dosages were available, the prevalence of persistent positivity (2 positive dosages spaced more than 12 weeks apart) was 21%.

Interestingly, a third of the cohort presented an antibody profile that did not allow them to be classified according to the classification criteria in force. This group corresponds to patients with a single positive dosage, either not recontrolled or recontrolled negative. This group was called Fluctuating. This fluctuating group was associated with arteriovenous fistula complications in a 2019 study.

Endothelial dysfunction is also implicated in the pathophysiology of APS. In clinical practice, the "flow mediated dilation" (FMD) test makes it possible to assess endothelial dysfunction in vivo. It involves the phenomenon of post-occlusive hyperemia which is mainly linked to NO and endothelium-dependent vasodilation. In the brachial artery, NO is the sole mediator of FMD. Endothelial dysfunction according to FMD has been described in populations with advanced chronic kidney disease, as well as patients with cardiovascular diseases. Hemodialysis patients with delayed/absence of arteriovenous fistula maturation have more pathological FMDs compared to dialysis patients without fistula problems. However, the additive role of aPL in this different population has not been studied in terms of endothelial dysfunction by FMD.

The objective of this study is to evaluate the weight of antiphospholipid biology on endothelial dysfunction in hemodialysis patients, using the FMD test.

1. Compare endothelial dysfunction by FMD according to the stage of chronic kidney disease and in comparison to a control group without chronic kidney disease.
2. Characterize the FMD pre or post dialysis and according to the duration of the long (for example between Thursday and Sunday) vs. short (between Tuesday and Thursday) inter-dialytic period.
3. Evaluate the relationship between endothelial dysfunction according to FMD, aPL positivity and arteriovenous fistula complications in hemodialysis patients.
4. Evaluate the risk factors associated with endothelial dysfunction according to FMD, and in particular evaluate the impact of antiphospholipid antibodies.
5. Evaluate the correlation between endothelial dysfunction according to FMD and other markers of endothelial dysfunction (urinary NO and metabolites of urinary NO, PGI2, endothelin, PGH2).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic kidney disease from stage G3a to G5
* Healthy volunteers

Exclusion Criteria:

* Patients with chronic kidney disease stage G5 with no dosage available of antiphospholipid antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Nitric oxide (NO) plasma level | pre-intervention
  Nitric oxide (NO) plasma level
Endothelin 1 (ET-1) plasma level | pre-intervention
  Endothelin 1 (ET-1) plasma level
E-Selectine plasma level | pre-intervention
  E-Selectine plasma level
P-Selectine plasma level | pre-intervention
  P-Selectine plasma level
Intercellular Adhesion Molecule 1 (ICAM-1) plasma level | pre-intervention
  Intercellular Adhesion Molecule 1 (ICAM-1) plasma level
Interleukin 6 (IL-6) plasma level | pre-intervention
  Interleukin 6 (IL-6) plasma level
Nitric oxide (NO) urine concentration | pre-intervention
  Nitric oxide (NO) urine concentration
Endothelin 1 (ET-1) urine concentration | pre-intervention
  Endothelin 1 (ET-1) urine concentration
Tumour Necrosis Factor alpha (TNF alpha) urine concentration | pre-intervention
  Tumour Necrosis Factor alpha (TNF alpha) urine concentration
Interleukin 6 (IL-6) urine concentration | pre-intervention
  Interleukin 6 (IL-6) urine concentration
Flow mediated dilatation test result (%) | pre-intervention
  Flow-mediated dilation (FMD) is a non-invasive vascular function test that measures the change in artery diameter in response to reactive hyperemia. The result of the test is expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Brugmann University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No